CLINICAL TRIAL: NCT00120289
Title: AIM HIGH: Niacin Plus Statin to Prevent Vascular Events
Brief Title: Niacin Plus Statin to Prevent Vascular Events
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: AIM-HIGH was stopped on the recommendation of the DSMB because of lack of efficacy of niacin in preventing primary outcome events.
Sponsor: Axio Research. LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Abbott (Industry)
Responsible Party: Principal Investigator, Ruth McBride, Co-Director, Coordinating Center, Axio Research. LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 226; U01HL081649 (NIH); U01HL081616 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-15 (Estimated); Results first posted 2015-06-17 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Cerebrovascular Accident; Coronary Disease; Atherosclerosis; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Stroke; Coronary Disease; Atherosclerosis; Myocardial Infarction | interventions — Niacin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Therapy (Experimental): Extended release niacin plus simvastatin
  Interventions: Drug: Extended release niacin; Drug: Simvastatin
- Monotherapy (Active Comparator): Simvastatin alone
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Extended release niacin — 2,000 mg/day or 1,500 mg/day if higher dose not tolerated
  Other Names: Niaspan
  Arms: Combination Therapy
Drug: Simvastatin — Dose adjusted to achieve LDL-C 40 mg/dL - 80 mg/dL, adding ezetimibe (10 mg/day) if needed to achieve LDL-C target
  Other Names: Zocor

SUMMARY:
The purpose of this study is to determine whether raising "good cholesterol" with a drug based on the vitamin niacin, while lowering "bad cholesterol" with a statin drug, can prevent more heart disease than the statin alone.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) remains the leading cause of death and disability in the Western world, with approximately 12.6 million individuals in the United States having a history of myocardial infarction (MI), angina, or both. There is mounting evidence that "conventional" therapies aimed at traditional risk factors have not optimized clinical outcomes. For example, in the Heart Protection Study with 20,536 subjects, the 5-year risk of a first major vascular event (nonfatal MI or CHD death, stroke, or coronary or noncoronary revascularization) among placebo-treated patients was 25%. Treatment with simvastatin reduced this risk to 20% over 5 years, which would project out to a 10-year risk of 40%. (The National Cholesterol Education Program Adult Treatment Panel III considers "high risk" or CHD equivalent a 10-year risk of an event greater than 20%.) Even among patients entering the study with baseline low density lipoprotein cholesterol (LDL-C) already near or at goal (i.e., LDL-C less than 116 mg/dL) and who achieved a mean on-trial LDL-C of 70 mg/dL with simvastatin, the 5-year risk of an event was still 18% (projecting to a 10-year risk of 36%). This residual and unacceptably high risk is likely due to the increasing prevalence of obesity, type II diabetes mellitus, and the metabolic syndrome. These disorders are typically accompanied by a constellation of abnormalities that include impaired glycemic control, hypertension, procoagulant and inflammatory states, and atherogenic dyslipidemia. The latter includes a wide spectrum of lipid abnormalities (low HDL-C, high triglycerides and triglyceride-rich remnant lipoproteins, and a preponderance of small dense, highly-oxidizable LDL particles).

Conventional LDL-C-focused therapies are not effective in targeting this type of dyslipidemia. Evidence that therapy directed at atherogenic dyslipidemia among patients with CHD can lower outcomes was shown with gemfibrozil in the VA-HIT trial, which showed a 22 to 24% cardiovascular (CV) event reduction by raising HDL-C (by an average of 6%) and lowering triglycerides (by an average of 31%). Niacin is an even more effective agent for simultaneously raising HDL-C and lowering triglycerides and levels of small dense LDL, and holds the most promise among existing therapies for substantial risk reduction in this population when added to a statin. This was demonstrated in the HDL Atherosclerosis Treatment Study (HATS) trial in which atherosclerosis progression was virtually halted and CV events were reduced by 60 to 90% using combined niacin plus statin therapy.

DESIGN NARRATIVE:

AIM-HIGH is a multicenter, randomized, double-blind, parallel-group, controlled clinical trial designed to test whether the drug combination of extended release niacin plus simvastatin is superior to simvastatin alone, at comparable levels of on-treatment LDL-C, for delaying the time to a first major CV disease outcome over a 4-year median follow-up in patients with atherogenic dyslipidemia. Prior clinical trials have found only 25 to 35% CV risk reduction using statin monotherapy (i.e., event rate 2/3 to 3/4 of placebo rate). The study is needed to confirm whether statin-niacin combination therapy, designed to target a wider spectrum of dyslipidemic factors in addition to LDL-C, will provide a more substantial (greater than 50%) reduction of CV events. Epidemiologic studies confirm the high prevalence of atherogenic dyslipidemia and its impact on CV event rates. Preliminary clinical trials suggest that targeting these factors with dyslipidemic therapy will reduce CV events. The study will enroll an estimated 3,300 men and women more than 45 years old at high risk of recurrent CV events by virtue of having established CV disease together with the two dyslipidemic elements of metabolic syndrome: low HDL-cholesterol (HDL-C) (less than or equal to 40 mg/dl) and high triglycerides (TG) (greater than or equal to 150 mg/dl). The study specifically aims to test this hypothesis for the primary composite clinical end point of CHD death, nonfatal MI, ischemic stroke, hospitalization for acute coronary syndrome with objective evidence of ischemia (troponin-positive or ST-segment deviation), or symptom-driven coronary or cerebral revascularization. Secondary end points include the composite of CHD death, nonfatal MI, ischemic stroke, or hospitalization for high-risk acute coronary syndrome; the composite of CHD death, nonfatal MI or ischemic stroke; and cardiovascular mortality.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 45 and older with established vascular disease and atherogenic dyslipidemia
* Established vascular disease defined as one or more of the following: (1) documented coronary artery disease (CAD); (2) documented cerebrovascular or carotid disease; (3) documented symptomatic peripheral arterial disease (PAD)
* Atherogenic dyslipidemia defined as: (1) LDL-C of less than or equal to 160 mg/dL (4.1 mmol/L); (2) HDL-C of less than or equal to 40 mg/dL (1.0 mmol/L) for men or less than or equal to 50 mg/dL (1.3 mmol/L) for women; (3) TG greater than or equal to 150 mg/dL (1.7 mmol/L) and less than or equal to 400 mg/dL (4.5 mmol/L)
* For patients entering the trial on a statin: (1) the upper limit for LDL-C is adjusted according to the specific statin and statin dose; (2) HDL-C of less than or equal to 42 mg/dL (1.1 mmol/L) for men or less than or equal to 53 mg/dL (1.4 mmol/L) for women; (3) TG greater than or equal to 125 mg/dL (1.4 mmol/L) and less than or equal to 400 mg/DL (4.5 mmol/L)

Exclusion Criteria:

* Coronary artery bypass graft (CABG) surgery within 1 year of planned enrollment (run-in phase)
* Percutaneous coronary intervention (PCI) within 4 weeks of planned enrollment (run-in phase)
* Hospitalization for acute coronary syndrome and discharge within 4 weeks of planned enrollment (run-in phase)
* Fasting glucose greater than 180 mg/dL (10 mmol/L) or hemoglobin A1C greater than 9%
* For patients with diabetes, inability or refusal to use a glucometer for home monitoring of blood glucose
* Concomitant use of drugs with a high probability of increasing the risk for hepatotoxicity or myopathy, such as those predominantly metabolized by cytochrome P450 system 3A4, including but not limited to cyclosporine, gemfibrozil, fenofibrate, itraconazole, ketoconazole, HIV protease inhibitors, nefazodone, verapamil, amiodarone; lipid-lowering drugs (other than the investigational drugs) such as statins, bile-acid sequestrants, cholesterol absorption inhibitors (e.g., ezetimibe), fibrates or high-dose, antioxidant vitamins (vitamins C, E, or beta carotene) that can interfere with the HDL-raising effect of niacin

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3414 (Actual)
Dates: Start 2005-09; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth McBride, Study Director — Axio Research Corporation; William E. Boden, MD, Principal Investigator — Samuel S. Stratton VA Medical Center; Jeffrey Probstfield, MD, Principal Investigator — University of Washington
Locations (91):
- United States (68):
  - Cardiovascular Associates, P.C., Birmingham, Alabama
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - Carl T. Hayden VAMC Phoenix Medical Service, Pheonix, Arizona
  - Cardiovascular Consultants Ltd, Phoenix, Arizona
  - Diabetes Center of Excellence, Phoenix, Arizona
  - Tucson Clinical Research (Eastside Site), Tucson, Arizona
  - Tucson Clinical Research (Northwest Site), Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center, Burbank, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - Christiana Care Health Services, Newark, Delaware
  - University of Miami, Miami, Florida
  - Heart & Vascular Research Center, Sarasota, Florida
  - James A. Haley Veteran's Hospital, Tampa, Florida
  - Idaho State University, Pocatello, Idaho
  - Parkview Research Center, Fort Wayne, Indiana
  - Iowa Heart Center, P.C., Des Moines, Iowa
  - Lipid Research Clinic, University of Iowa, Iowa City, Iowa
  - Maine Center for Lipids & Cardiovascular Health, Scarborough, Maine
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - Veterans Affairs Health System of Ann Arbor, Michigan, Ann Arbor, Michigan
  - Grunberger Diabetes Institute, Bloomfield Hills, Michigan
  - Berman Center for Outcomes and Clinical Research, Minneapolis, Minnesota
  - HealthPartners Riverside Clinic, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Phalen Village Clinic, Saint Paul, Minnesota
  - University of Minnesota, Twin Cities, Minnesota
  - G.V. (Sonny) Montgomery VAMC, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - Alegent Health Heart & Vascular Specialists, Papillion, Nebraska
  - Cooper Clinical Trials Center, Cherry Hill, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - UMDNJ -Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New Mexico VA Healthcare Systems, Albuquerque, New Mexico
  - Kaleida Health/Diabetes Center, Buffalo, New York
  - Mid Valley Cardiology, Kingston, New York
  - VA New York Harbor Healthcare System, New York, New York
  - Columbia University, New York, New York
  - Syracuse Preventive Cardiology, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University - Geriatrics/Gerontology, Greensboro, North Carolina
  - Wake Forest University Health Sciences - Department of Cardiology, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine - Internal Medicine/Endocrinology, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - St Vincent Charity Hospital - The Center for Vascular Health, Cleveland, Ohio
  - North Ohio Research, Ltd., Sandusky, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Cardiology Associates, Philadelphia, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Women's Cardiac Center at The Miriam Hospital, Providence, Rhode Island
  - Internal Medicine Associates of Greenville, Greenville, South Carolina
  - VAMC Memphis - Hypertension/Lipid Research Clinic, Memphis, Tennessee
  - Kelsey Research Foundation, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia - UVA Cardiology, Charlottesville, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - University of Washington, Northwest Lipid Research Center, Seattle, Washington
  - University of Washington, Coronary Atherosclerosis Research Lab, Seattle, Washington
  - VA Cardiology Research, Seattle, Washington
  - Washington State University, Spokane, Washington
  - CARE Foundation, Inc., Wausau, Wisconsin
- Canada (23):
  - Heart Health Institute, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver Hospital, Vancouver, British Columbia
  - Victoria Heart Institute, Victoria, British Columbia
  - Health Sciences Center, Diabetes Research Group, Winnipeg, Manitoba
  - New Brunswick Heart Center, Saint John, New Brunswick
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Cardiology Associates VRH, Kentville, Nova Scotia
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - McConnell Medical Center, Cornwall, Ontario
  - Sudbury Cardiovascular Research, Greater Sudbury, Ontario
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - LHSC University Hospital, London, Ontario
  - Newmarket Cardiology Research Group, Newmarket, Ontario
  - St. Michael's Hospital Health Centre, Toronto, Ontario
  - Clinique de Cardiologie de Lévis, Lévis, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Recherches Clinicar, Québec, Quebec
  - Clinique des maladies lipidiques de Québec, Québec, Quebec
  - CSSS Beauce, St-Georges de Beauce, Quebec
  - CSSS du Sud de Lanaudière - Hôpital Pierre-Le Gardeur, Terrebonne, Quebec

REFERENCES:
- [Background] AIM-HIGH Investigators. The role of niacin in raising high-density lipoprotein cholesterol to reduce cardiovascular events in patients with atherosclerotic cardiovascular disease and optimally treated low-density lipoprotein cholesterol: baseline characteristics of study participants. The Atherothrombosis Intervention in Metabolic syndrome with low HDL/high triglycerides: impact on Global Health outcomes (AIM-HIGH) trial. Am Heart J. 2011 Mar;161(3):538-43. doi: 10.1016/j.ahj.2010.12.007. Epub 2011 Feb 2. PMID 21392609
- [Background] AIM-HIGH Investigators. The role of niacin in raising high-density lipoprotein cholesterol to reduce cardiovascular events in patients with atherosclerotic cardiovascular disease and optimally treated low-density lipoprotein cholesterol Rationale and study design. The Atherothrombosis Intervention in Metabolic syndrome with low HDL/high triglycerides: Impact on Global Health outcomes (AIM-HIGH). Am Heart J. 2011 Mar;161(3):471-477.e2. doi: 10.1016/j.ahj.2010.11.017. Epub 2011 Feb 2. PMID 21392600
- [Result] AIM-HIGH Investigators; Boden WE, Probstfield JL, Anderson T, Chaitman BR, Desvignes-Nickens P, Koprowicz K, McBride R, Teo K, Weintraub W. Niacin in patients with low HDL cholesterol levels receiving intensive statin therapy. N Engl J Med. 2011 Dec 15;365(24):2255-67. doi: 10.1056/NEJMoa1107579. Epub 2011 Nov 15. PMID 22085343
- [Result] Teo KK, Goldstein LB, Chaitman BR, Grant S, Weintraub WS, Anderson DC, Sila CA, Cruz-Flores S, Padley RJ, Kostuk WJ, Boden WE; AIM-HIGH Investigators. Extended-release niacin therapy and risk of ischemic stroke in patients with cardiovascular disease: the Atherothrombosis Intervention in Metabolic Syndrome with low HDL/High Triglycerides: Impact on Global Health Outcome (AIM-HIGH) trial. Stroke. 2013 Oct;44(10):2688-93. doi: 10.1161/STROKEAHA.113.001529. Epub 2013 Jul 23. PMID 23881958
- [Result] Albers JJ, Slee A, O'Brien KD, Robinson JG, Kashyap ML, Kwiterovich PO Jr, Xu P, Marcovina SM. Relationship of apolipoproteins A-1 and B, and lipoprotein(a) to cardiovascular outcomes: the AIM-HIGH trial (Atherothrombosis Intervention in Metabolic Syndrome with Low HDL/High Triglyceride and Impact on Global Health Outcomes). J Am Coll Cardiol. 2013 Oct 22;62(17):1575-9. doi: 10.1016/j.jacc.2013.06.051. Epub 2013 Aug 21. PMID 23973688
- [Result] Guyton JR, Slee AE, Anderson T, Fleg JL, Goldberg RB, Kashyap ML, Marcovina SM, Nash SD, O'Brien KD, Weintraub WS, Xu P, Zhao XQ, Boden WE. Relationship of lipoproteins to cardiovascular events: the AIM-HIGH Trial (Atherothrombosis Intervention in Metabolic Syndrome With Low HDL/High Triglycerides and Impact on Global Health Outcomes). J Am Coll Cardiol. 2013 Oct 22;62(17):1580-4. doi: 10.1016/j.jacc.2013.07.023. Epub 2013 Jul 31. PMID 23916935
- [Derived] Ronsein GE, Vaisar T, Davidson WS, Bornfeldt KE, Probstfield JL, O'Brien KD, Zhao XQ, Heinecke JW. Niacin Increases Atherogenic Proteins in High-Density Lipoprotein of Statin-Treated Subjects. Arterioscler Thromb Vasc Biol. 2021 Aug;41(8):2330-2341. doi: 10.1161/ATVBAHA.121.316278. Epub 2021 Jun 17. PMID 34134520
- [Derived] Tuteja S, Qu L, Vujkovic M, Dunbar RL, Chen J, DerOhannessian S, Rader DJ. Genetic Variants Associated With Plasma Lipids Are Associated With the Lipid Response to Niacin. J Am Heart Assoc. 2018 Oct 2;7(19):e03488. doi: 10.1161/JAHA.117.008461. PMID 30371334
- [Derived] Toth PP, Jones SR, Slee A, Fleg J, Marcovina SM, Lacy M, McBride R, Boden WE. Relationship between lipoprotein subfraction cholesterol and residual risk for cardiovascular outcomes: A post hoc analysis of the AIM-HIGH trial. J Clin Lipidol. 2018 May-Jun;12(3):741-747.e11. doi: 10.1016/j.jacl.2018.03.077. Epub 2018 Mar 9. PMID 29627296
- [Derived] O'Brien KD, Hippe DS, Chen H, Neradilek MB, Probstfield JL, Peck S, Isquith DA, Canton G, Yuan C, Polissar NL, Zhao XQ, Kerwin WS. Longer duration of statin therapy is associated with decreased carotid plaque vascularity by magnetic resonance imaging. Atherosclerosis. 2016 Feb;245:74-81. doi: 10.1016/j.atherosclerosis.2015.11.032. Epub 2015 Dec 1. PMID 26708287
- See also: AIM-HIGH Web site for patients — http://www.aimhigh-heart.com/
- Available data/document: Individual Participant Data Set: AIM-HIGH — http://biolincc.nhlbi.nih.gov/studies/aimhigh/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol: AIM-HIGH — http://biolincc.nhlbi.nih.gov/studies/aimhigh/
- Available data/document: Study forms: AIM-HIGH — http://biolincc.nhlbi.nih.gov/studies/aimhigh/

RESULTS

PARTICIPANT FLOW:
Groups:
- ERN + Simvastatin: Extended release niacin plus simvastatin
  Extended release niacin: 2,000 mg/day or 1,500 mg/day if higher dose not tolerated
  Simvastatin: Dose adjusted to achieve LDL-C 40 mg/dL - 80 mg/dL, adding ezetimibe (10 mg/day) if needed to achieve LDL-C target
- Placebo + Simvastatin: Simvastatin alone
  Simvastatin: Dose adjusted to achieve LDL-C 40 mg/dL - 80 mg/dL, adding ezetimibe (10 mg/day) if needed to achieve LDL-C target
Period: Overall Study
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Started | 1718 | 1696
Completed | 1597 | 1587
Not Completed | 121 | 109
Not completed — Death | 96 | 82
Not completed — Lost to Follow-up | 11 | 14
Not completed — Withdrawal by Subject | 14 | 13

BASELINE CHARACTERISTICS:
Population: Intention-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin | Total
Number analyzed (Participants) | 1718 | 1696 | 3414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 917 | 915 | 1832
  >=65 years | 801 | 781 | 1582
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.8) | 63.7 (8.7) | 63.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 251 | 504
  Male | 1465 | 1445 | 2910
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 77 | 140
  Not Hispanic or Latino | 1654 | 1619 | 3273
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 11 | 22
  Asian | 20 | 21 | 41
  Native Hawaiian or Other Pacific Islander | 7 | 5 | 12
  Black or African American | 68 | 49 | 117
  White | 1572 | 1576 | 3148
  More than one race | 40 | 33 | 73
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1179 | 1167 | 2346
  Canada | 539 | 529 | 1068
Lipids and Lipoproteins at Baseline [Mean (Standard Deviation); unit: mg/dL]
  LDL-C | 74.2 (23.4) | 74.0 (22.7) | 74.1 (23)
  HDL-C | 34.5 (5.6) | 34.9 (5.6) | 34.7 (5.6)
  Triglycerides | 183.5 (66.7) | 181.9 (66.9) | 182.7 (66.8)
  non-HDL cholesterol | 110.8 (27.5) | 110.3 (26) | 110.6 (26.8)
  HDL2-C | 6 (2.3) | 6.2 (2.4) | 6.1 (2.3)
  HDL3-C | 28.5 (4.2) | 28.7 (4.1) | 28.6 (4.1)
  Apolipoprotein A-I | 122.4 (16.2) | 123.7 (16.3) | 123.1 (16.2)
  Apolipoprotein B | 83.2 (20.2) | 82.9 (20.7) | 83 (20.4)
  Lipoprotein (a) | 77.3 (87.8) | 75.5 (89.6) | 76.4 (88.7)
Clinical History [Number; unit: participants]
  History of myocardial infarction (MI) | 968 | 955 | 1923
  History of CABG | 600 | 627 | 1227
  History of Percutaneous Coronary Intervention | 1057 | 1044 | 2101
  History of stroke or cerebrovascular disease | 358 | 362 | 720
  History of peripheral vascular disease | 234 | 231 | 465
  Metabolic syndrome | 1414 | 1353 | 2767
  History of diabetes (Type 1 or 2) | 588 | 570 | 1158
Concomitant Medications at Baseline [Number; unit: participants]
  Statins | 1595 | 1601 | 3196
  Beta-blockers | 1377 | 1342 | 2719
  ACE inhibitor or Angiotensin Receptor Blocker | 1258 | 1271 | 2529
  Aspirin or other antiplatelet or anticoagulant | 1680 | 1654 | 3334

OUTCOME MEASURES:

1. Primary Outcome: Composite End Point of CHD Death, Nonfatal MI, Ischemic Stroke, Hospitalization for Non-ST Segment Elevation Acute Coronary Syndrome (ACS), or Symptom-driven Coronary or Cerebral Revascularization
Time Frame: Time to first event measured from date of randomization through last follow-up visit (common termination) for an average of 36 months follow-up, maximum 66 months.
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Number analyzed (Participants) | 1718 | 1696
participants | 282 | 274
Statistical Analysis 1: Comparison: ERN + Simvastatin vs Placebo + Simvastatin; Test type: Superiority or Other; p = 0.80, Regression, Cox; Adjusting for gender and history of diabetes (randomization stratification factors); Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.87 to 1.21]

2. Secondary Outcome: Composite Endpoint of CHD Death, Non-fatal MI, High-risk ACS or Ischemic Stroke
Time Frame: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Number analyzed (Participants) | 1718 | 1696
participants | 171 | 158
Statistical Analysis 1: Comparison: ERN + Simvastatin vs Placebo + Simvastatin; Test type: Superiority or Other; p = .49, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.87 to 1.34]

3. Secondary Outcome: Composite Endpoint of CHD Death, Non-fatal MI, or Ischemic Stroke
Time Frame: as for outcome 1
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Number analyzed (Participants) | 1718 | 1696
participants | 156 | 138
Statistical Analysis 1: Comparison: ERN + Simvastatin vs Placebo + Simvastatin; Test type: Superiority or Other; p = .30, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.90 to 1.42]

4. Secondary Outcome: Cardiovascular Mortality
Time Frame: Time to first event measured from date of randomization through last follow-up visit (common termination), for an average of 36 months follow-up, maximum 66 months.
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Number analyzed (Participants) | 1718 | 1696
participants | 45 | 38
Statistical Analysis 1: Comparison: ERN + Simvastatin vs Placebo + Simvastatin; Test type: Superiority or Other; p = 0.47, Regression, Cox; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.76 to 1.80]

ADVERSE EVENTS:
Time Frame: Randomization through final study visit after recommendation to curtail study (June - September 2011)
Arm/Group | ERN + Simvastatin | Placebo + Simvastatin
Serious Adverse Events (participants affected / at risk) | 587/1718 | 551/1696
Other Adverse Events (participants affected / at risk) | 1413/1718 | 1345/1696
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ERN + Simvastatin (N=1718) | Placebo + Simvastatin (N=1696)
Anaemia (Blood and lymphatic system disorders) | 17 | 10
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Acute myocardial infarction (Cardiac disorders) | 3 | 3
Acute pulmonary oedema (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 16 | 21
Angina unstable (Cardiac disorders) | 6 | 5
Aortic valve calcification (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 27 | 25
Atrial flutter (Cardiac disorders) | 5 | 5
Atrial tachycardia (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 1
Atrioventricular block third degree (Cardiac disorders) | 2 | 4
Bradycardia (Cardiac disorders) | 2 | 8
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 10 | 9
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 21 | 30
Cardiomyopathy (Cardiac disorders) | 1 | 2
Chest discomfort (Cardiac disorders) | 5 | 7
Chest pain (Cardiac disorders) | 43 | 57
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 5 | 1
Cyanosis (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Dyspnoea (Cardiac disorders) | 31 | 38
Dyspnoea exertional (Cardiac disorders) | 1 | 5
Dyspnoea paroxysmal nocturnal (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 2
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 3 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 7
Presyncope (Cardiac disorders) | 2 | 4
Pulmonary oedema (Cardiac disorders) | 3 | 4
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 3 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1
Subvalvular aortic stenosis (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Syncope (Cardiac disorders) | 21 | 19
Tachycardia (Cardiac disorders) | 3 | 2
Tachycardia paroxysmal (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 6 | 5
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Hypospadias (Congenital, familial and genetic disorders) | 1 | 0
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Chorioretinal atrophy (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 1
Eye inflammation (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 22 | 10
Abdominal pain lower (Gastrointestinal disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 8 | 6
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 2
Colonic fistula (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 6
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulitis oesophageal (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 4 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 4 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 13
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 5
Haematochezia (Gastrointestinal disorders) | 3 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 3
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 12 | 7
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 2 | 2
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 11 | 3
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 5 | 4
Umbilical hernia (Gastrointestinal disorders) | 0 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Volvulus (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 20 | 9
Abasia (General disorders) | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 10 | 8
Chest discomfort (General disorders) | 2 | 6
Chest pain (General disorders) | 2 | 0
Chills (General disorders) | 1 | 2
Cyst (General disorders) | 1 | 0
Death (General disorders) | 3 | 1
Face oedema (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 11 | 6
Feeling abnormal (General disorders) | 1 | 0
Gait disturbance (General disorders) | 3 | 3
General physical health deterioration (General disorders) | 1 | 1
Hernia (General disorders) | 1 | 2
Hyperthermia (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Mass (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 12 | 18
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 4 | 5
Pain (General disorders) | 3 | 1
Pyrexia (General disorders) | 6 | 8
Sudden death (General disorders) | 1 | 0
Thirst (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 4
Cholecystitis acute (Hepatobiliary disorders) | 6 | 2
Cholelithiasis (Hepatobiliary disorders) | 8 | 7
Gallbladder pain (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Abscess neck (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 8 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 2 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 7 | 1
Bronchitis acute (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 26 | 13
Clostridium difficile colitis (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 6 | 4
Endocarditis (Infections and infestations) | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 2
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 4 | 2
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 0 | 1
Infected insect bite (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 4 | 0
Localised infection (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 4 | 4
Perianal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 38 | 27
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Postoperative infection (Infections and infestations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 0 | 3
Pyelonephritis (Infections and infestations) | 1 | 2
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 10
Septic embolus (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Sweat gland infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 19 | 10
Urosepsis (Infections and infestations) | 5 | 2
Wound infection (Infections and infestations) | 0 | 3
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 9
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Fracture of penis (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 2 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 6
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incision site complication (Injury, poisoning and procedural complications) | 2 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Injury asphyxiation (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 3
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 2
Narcotic intoxication (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pharyngeal injury (Injury, poisoning and procedural complications) | 0 | 1
Polytraumatism (Injury, poisoning and procedural complications) | 1 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 2
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 3
Wound decomposition (Injury, poisoning and procedural complications) | 0 | 1
Arteriogram coronary (Investigations) | 0 | 1
Arteriogram coronary normal (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 2 | 2
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 3
Cardiac stress test abnormal (Investigations) | 1 | 0
Ejection fraction abnormal (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 1
Haematocrit decreased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 2 | 2
Heart rate decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 2 | 1
Hepatic enzyme increased (Investigations) | 3 | 0
International normalised ratio increased (Investigations) | 1 | 1
Intraocular pressure increased (Investigations) | 0 | 1
Oxygen consumption increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 3 | 0
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic ulcer (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 3
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 6 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Oral intake reduced (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 18
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 24 | 28
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Benign neoplasm of ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the caecum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 14
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer stage IIIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 10
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 4
Coordination abnormal (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 2 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 21 | 19
Drooling (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 2
Essential tremor (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 0 | 3
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 4
Hemiparesis (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 5 | 2
Intracranial aneurysm (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 4 | 4
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 2
Migraine with aura (Nervous system disorders) | 0 | 1
Myelitis transverse (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Neuritis (Nervous system disorders) | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 5
Paresis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 2 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 1
Radicular pain (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 5 | 6
Tremor (Nervous system disorders) | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anger (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 7 | 8
Delirium (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 4 | 5
Depression suicidal (Psychiatric disorders) | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Dysphasia (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 1
Impaired self-care (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 3
Panic attack (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 4 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 4
Calculus urinary (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 2
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 6
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 4 | 7
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 7 | 4
Renal failure acute (Renal and urinary disorders) | 18 | 15
Renal failure chronic (Renal and urinary disorders) | 3 | 3
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urethral perforation (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 4 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 3
Breast cancer in situ (Reproductive system and breast disorders) | 1 | 0
Endometrial cancer recurrent (Reproductive system and breast disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 4
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 2
Cardioversion (Surgical and medical procedures) | 1 | 1
Coronary revascularisation (Surgical and medical procedures) | 1 | 0
Hypotensive anaesthesia procedure (Surgical and medical procedures) | 0 | 1
Peripheral revascularisation (Surgical and medical procedures) | 0 | 1
Shoulder arthroplasty (Surgical and medical procedures) | 1 | 0
Spinal decompression (Surgical and medical procedures) | 1 | 0
Stent placement (Surgical and medical procedures) | 1 | 1
Therapeutic embolisation (Surgical and medical procedures) | 1 | 0
Toe amputation (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 8 | 11
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 3
Aorto-duodenal fistula (Vascular disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Carotid artery aneurysm (Vascular disorders) | 0 | 1
Carotid artery disease (Vascular disorders) | 0 | 1
Carotid artery stenosis (Vascular disorders) | 1 | 2
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 9 | 6
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 2
Hypertension (Vascular disorders) | 5 | 5
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 11 | 8
Iliac artery stenosis (Vascular disorders) | 0 | 2
Intermittent claudication (Vascular disorders) | 2 | 4
Orthostatic hypotension (Vascular disorders) | 2 | 3
Peripheral artery aneurysm (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 3 | 3
Pulmonary embolism (Vascular disorders) | 4 | 5
Pulmonary hypertension (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Vascular pseudoaneurysm (Vascular disorders) | 5 | 1
Vasospasm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ERN + Simvastatin (N=1718) | Placebo + Simvastatin (N=1696)
Anaemia (Blood and lymphatic system disorders) | 41 | 34
Angina pectoris (Cardiac disorders) | 43 | 46
Atrial fibrillation (Cardiac disorders) | 43 | 30
Chest pain (Cardiac disorders) | 112 | 95
Dyspnoea (Cardiac disorders) | 89 | 89
Dyspnoea exertional (Cardiac disorders) | 26 | 40
Cataract (Eye disorders) | 80 | 77
Abdominal pain (Gastrointestinal disorders) | 39 | 34
Diarrhoea (Gastrointestinal disorders) | 136 | 63
Nausea (Gastrointestinal disorders) | 55 | 40
Vomiting (Gastrointestinal disorders) | 46 | 28
Fatigue (General disorders) | 87 | 74
Non-cardiac chest pain (General disorders) | 27 | 42
Oedema peripheral (General disorders) | 66 | 73
Bronchitis (Infections and infestations) | 82 | 68
Cellulitis (Infections and infestations) | 36 | 30
Herpes zoster (Infections and infestations) | 53 | 29
Influenza (Infections and infestations) | 61 | 62
Nasopharyngitis (Infections and infestations) | 113 | 121
Pneumonia (Infections and infestations) | 38 | 52
Sinusitis (Infections and infestations) | 80 | 71
Upper respiratory tract infection (Infections and infestations) | 72 | 59
Urinary tract infection (Infections and infestations) | 60 | 53
Contusion (Injury, poisoning and procedural complications) | 29 | 36
Blood glucose increased (Investigations) | 112 | 78
Diabetes mellitus (Metabolism and nutrition disorders) | 67 | 41
Gout (Metabolism and nutrition disorders) | 66 | 65
Arthralgia (Musculoskeletal and connective tissue disorders) | 138 | 158
Back pain (Musculoskeletal and connective tissue disorders) | 120 | 122
Muscle spasms (Musculoskeletal and connective tissue disorders) | 46 | 51
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 75 | 88
Myalgia (Musculoskeletal and connective tissue disorders) | 53 | 53
Neck pain (Musculoskeletal and connective tissue disorders) | 38 | 35
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 47 | 50
Pain in extremity (Musculoskeletal and connective tissue disorders) | 134 | 147
Dizziness (Nervous system disorders) | 95 | 122
Headache (Nervous system disorders) | 61 | 51
Hypoaesthesia (Nervous system disorders) | 36 | 35
Cough (Respiratory, thoracic and mediastinal disorders) | 57 | 52
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 27
Rash (Skin and subcutaneous tissue disorders) | 58 | 38
Hypertension (Vascular disorders) | 59 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No